CLINICAL TRIAL: NCT01655082
Title: Nicotine Patch Safety Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V00116 TD 2 02; 2011-005911-94 (EudraCT Number)
Record Dates: First submitted 2012-07-30; First posted 2012-08-01 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Smokers
Keywords: Smoking cessation; Nicotine; Tobacco Use Disorder; Central Nervous System Agents
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder | interventions — Tobacco Use Cessation Devices

ARMS (2):
- V0116 (Experimental): One patch per day (during 24 hours) for 21 days
  Interventions: Drug: V0116 transdermal patch
- Reference (Active Comparator): One patch per day (during 24 hours) for 21 days
  Interventions: Drug: Nicotine transdermal patch

INTERVENTIONS:
Drug: V0116 transdermal patch — One patch per day (during 24 hours) for 21 days
  Arms: V0116
Drug: Nicotine transdermal patch — One patch per day (during 24 hours) for 21 days
  Arms: Reference

SUMMARY:
The purpose of this study is to evaluate the safety profile of a repeated application of a new transdermal patch compared to a reference product during 3 weeks, in a large population.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged more than 18 years
* Regular smoker motivated to stop tobacco consumption
* Current smoker of > or = 20 cigarettes/day and < or = 25 cigarettes/day or Fagerström score > or = 5 (for smokers between 10 to 20 cigarettes/day)

Exclusion Criteria:

* Any visible skin disorder, abnormal skin pigmentation or other dermatologic disease which, in the opinion of the investigator would interfere with the assessment of the different parameters
* Current or past serious chronic cardiovascular, renal, hepatic, gastrointestinal (including duodenal or gastric ulcer), endocrine, hematological, neuropsychiatric, immunosuppressive condition or allergic disease, myopathies, epileptic seizures, bleeding tendency, cancer
* History of angina pectoris, myocardial infarction or stroke in the previous 3 months, coronary artery vasospasm, cardiac arrhythmia, acute stroke
* Clinically relevant abnormal findings on the physical examination (e.g large scars on the application zone)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2012-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Safety | up to Day 22
  Evaluation of local safety (number of subjects with skin irritation / number of subjects by score of adhesiveness) and general safety (number of subjects with emergent adverse events or changes from baseline to end of study in vital signs, electrocardiogram and clinical laboratory parameters).

SECONDARY OUTCOMES:
Sensory profile | Day 22
  Visual Analogic Scales (sensations linked to patch application and removal)
Global assessment by the patient | Day 22
  Visual Analog Scale Scale and questionnaires
Subject behaviours | up to Day 22
  nicotine consumption

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Gières
  - Pierre-Bénite
  - Rennes
  - Rueil-Malmaison